CLINICAL TRIAL: NCT05949086
Title: An Online Evaluation of Work Chat: A Virtual Workday Among Employed Autistic Adults
Brief Title: An Online Evaluation of Work Chat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); SIMmersion, LLC (Industry)
Responsible Party: Principal Investigator, Matthew Smith, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HUM00228606; R44MH123359-01 (NIH)
Record Dates: First submitted 2023-07-07; First posted 2023-07-17 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Work Chat Later (No Intervention): This group will not receive Work Chat during the study, but will receive Work Chat access after data collection is complete.
- Work Chat Now (Experimental): Behavioral: Work Chat: An Interactive Virtual Workday Work Chat will be a simulation training using virtual characters to role-play conversations. It will contain conversations with a coworker, a customer, and a supervisor within a workplace setting.
  Interventions: Behavioral: Work Chat

INTERVENTIONS:
Behavioral: Work Chat — Work Chat will be a simulation training using virtual characters to role-play conversations. It will contain conversations with a coworker, a customer, and a supervisor within a workplace setting.
  Arms: Work Chat Now

SUMMARY:
This study is aiming to see if it is feasible for the intervention Work Chat to be delivered in a completely online setting to adults with autism spectrum disorder.

DETAILED DESCRIPTION:
Nearly 50,000 youth with autism spectrum disorder (ASD) transition from high school to adult life each year, with only 25% of these transition-age youth with ASD (TAY-ASD) getting jobs within 2 years of graduation. TAY-ASD's ability to sustain employment is even more challenging due in part to their social cognitive deficits (e.g., poorly reading social cues) that disrupt communicating with customers, coworkers, and supervisors. Research shows nearly 90% of job dismissals among TAY-ASD are attributed to poor work-based social functioning (e.g., poorly communicating with upset customers). The subsequent unemployment has damaging effects on their mental, physical, and economic health. A critical gap in federally-mandated services to support youth with ASD as they transition from school-to-adult life is the lack of evidence-based practice to enhance their work-based social functioning. Given that TAY-ASD report computerized training tools are highly acceptable and improve their real-world outcomes, the investigators propose to address this critical barrier to sustained employment by developing and evaluating a novel and scalable computerized training tool to enhance their conversations with customers, coworkers and supervisors at work.

The investigators are aiming to see if it is feasible for Work Chat to be delivered in a completely online setting and not within schools or other sites. The investigators are also evaluating the tool specifically with employed adults who have autism spectrum disorder.

ELIGIBILITY:
Inclusion Criteria:

* Autism Spectrum Disorder
* 18 years or older
* Has 4th grade or higher reading level
* Employed or Unemployed and searching for employment within the next 3 months
* Has access to a computer, laptop, or tablet that has connection to the internet and a camera (not including smartphone)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2023-07-07 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Change in Theory of Mind - Hinting Task | Baseline and posttest (approximately 6 weeks after baseline)
  Measured by the hinting task (Corcoran, Mercer, & Frith, 1995), which comprises 10 short stories describing an interaction between two characters, all of which end with one of the characters making a hint. At the end of each passage, the participant is asked what the hint meant. If they give a correct response (score 2), they move onto the next item. If they fail, they are provided with extra information to help interpret the hint. A correct recognition of the hint at this stage scores 1. Total score can be 0-20, with a higher score being a better outcome.
Change in Emotion Recognition Ability - MiniPONs | Baseline and posttest (approximately 6 weeks after baseline)
  Measured by the MiniPONS, which is a short, multichannel version of the established Profile of Nonverbal Sensitivity (PONS) test (Rosenthal et al., 1979). The short multichannel version (64 items) available here correlates very highly with the full version and shows reasonable construct validity through significant correlations with other tests of emotion recognition ability. A total score is calculated at the end, total score can be 0-64, with a higher score being a better outcome.
Greater sustained employment by 9 Months | 9 Month Follow Up (approximately 9 Months after randomization)
  Self-report employment surveys completed at baseline and follow ups. Employment will be tracked as 0 (no job) and 1 (job). Higher scores indicate a better outcome.
Change in Managing Emotions | Baseline and posttest (approximately 6 weeks after baseline)
  The Mayer-Salovey-Caruso Emotional Intelligence Test (MSCEIT) is an ability-based test designed to measure the four branches of the EI model of Mayer and Salovey. This study will only use the Managing Emotions Subscale, which measures the ability to be be open to emotions and feelings and integrate emotions with thinking. There are 29 scenarios presented, with higher score ranges indicating a positive outcome and lower score ranges indicating a worse outcome. The score ranges are as follows: Improve (worse), Consider Developing, Competent, Skilled, and Expert (positive).

SECONDARY OUTCOMES:
Change in Anxiety | Baseline and posttest (approximately 6 weeks after baseline)
  Measured by the Social Interaction Anxiety Scale (SIAS) self-report survey. Items are on a 5 point scale with 0 being "not at all" and 4 being "extremely". Total score can be 0-80, with higher scores indicating higher anxiety, a worse outcome.

OTHER OUTCOMES:
Change in Social Competence/Applied Social Ability | Baseline and posttest (approximately 6 weeks after baseline)
  Measured by Social Skills Performance Assessment (SSPA). Roleplay performance: The SSPA includes two brief (3-minute) roleplays in which participants engage in a conversation with an unknown confederate who plays the role of a new neighbor(NN) or a landlord (LL). The NN and LL role plays were video recorded at the pre- and posttest visits and were blindly rated by use of an anchoring system. The NN roleplay was scored on eight items via a 5-point scale (e.g., 5,very interested, to 1, very disinterested), and the LL roleplay was scored on nine items via a 5-point scale (e.g., 5,very focused, to 1, very unfocused). The two role-play scores were combined to create one total pretest score and one total posttest score. Sum scores could have a minimum of 17 and maximum of 85. Higher scores indicated better skills.
Change in Interpersonal Communication at Work | Baseline and posttest (approximately 6 weeks after baseline) and 3-month, 6-month, 9-month follow up after randomization.
  Measured by the Interpersonal Communication at Work Scale. There are 4 items on a scale from 1 (Less than once per month or never) to 5 (several times per day). A higher score indicates a more negative outcome.
Change in Job Satisfaction | Baseline and posttest (approximately 6 weeks after baseline) and 3-month, 6-month, 9-month follow up after randomization.
  Measured by the Job Satisfaction of Persons with Disability Scale. There are 14 items on a scale from 1 Strongly Disagree to 7 Strongly Agree with a higher score indicating a more positive score. Total scores can range from 14-98.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Smith, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-11-12): https://cdn.clinicaltrials.gov/large-docs/86/NCT05949086/ICF_000.pdf